CLINICAL TRIAL: NCT00352079
Title: A Phase III Study of IRESSA in Combination With Intravesical BCG Versus Intravesical BCG Alone in High Risk Superficial Transitional Cell Carcinoma of the Bladder
Brief Title: BCG With or Without Gefitinib in Treating Patients With High-Risk Bladder Cancer
Status: Terminated | Phase: Phase 3 | Type: Interventional
Why Stopped: terminated due to poor accrual
Sponsor: NCIC Clinical Trials Group (Network)
Responsible Party: Sponsor
Organization: Canadian Cancer Trials Group (Network)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: BL11; CAN-NCIC-BL11 (Other: PDQ); CDR0000486873 (Other: PDQ)
Record Dates: First submitted 2006-07-13; First posted 2006-07-14 (Estimated); Last update posted 2023-08-04 (Actual); Status verified 2020-04

CONDITIONS: Bladder Cancer
Keywords: transitional cell carcinoma of the bladder; stage 0 bladder cancer; stage I bladder cancer; recurrent bladder cancer
MeSH Terms: conditions — Urinary Bladder Neoplasms | interventions — BCG Vaccine; Gefitinib

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intravesicle BCG (Active Comparator): Induction:
  q weekly x 6 (cycle 1)
  Maintenance:
  q weekly x 3 at 3, 6, 12, 18, 24, 30, 36 months postrandomization (cycles 2 - 8)
  Interventions: Biological: BCG vaccine; Procedure: quality-of-life assessment
- Iressa and Intravesicle BCG (Active Comparator): Intravesical BCG:
  Induction:
  q weekly x 6 (cycle 1)
  Maintenance:
  q weekly x 3 at 3, 6, 12, 18, 24, 30, 36 months post- 2 randomization (cycles 2 - 8)
  Iressa® 250 mg PO Daily for 12 weeks starting on day 1 of each cycle of intravesical BCG therapy (cycles 1 - 8)
  Interventions: Biological: BCG vaccine; Drug: gefitinib; Procedure: quality-of-life assessment

INTERVENTIONS:
Biological: BCG vaccine — Intravesical BCG:
  Induction:
  q weekly x 6 (cycle 1)
  Maintenance:
  q weekly x 3 at 3, 6, 12, 18, 24, 30, 36 months post- 2 randomization (cycles 2 - 8)
Drug: gefitinib — Iressa® 250 mg PO Daily for 12 weeks starting on day 1 of each cycle of intravesical BCG therapy (cycles 1 - 8)
  Arms: Iressa and Intravesicle BCG
Procedure: quality-of-life assessment — Each cycle and at 3 and 6 months after treatment discontinuation

SUMMARY:
RATIONALE: Biological therapies, such as BCG, may stimulate the immune system in different ways and stop tumor cells from growing. Gefitinib may stop the growth of tumor cells by blocking some of the enzymes needed for cell growth. Giving BCG together with gefitinib may kill more tumor cells. It is not yet known whether BCG is more effective with or without gefitinib in treating bladder cancer.

PURPOSE: This randomized phase III trial is studying BCG and gefitinib to see how well they work compared to BCG alone in treating patients with high-risk bladder cancer.

DETAILED DESCRIPTION:
OBJECTIVES:

Primary

* Compare the impact of gefitinib and intravesical BCG vs intravesical BCG alone on time to treatment failure in patients with high-risk, superficial transitional cell carcinoma of the bladder.

Secondary

* Compare the complete response rates in patients with carcinoma in situ receiving gefitinib and intravesical BCG vs patients receiving intravesical BCG alone.
* Compare the time to recurrence in patients treated with these regimens.
* Compare the time to progression in patients treated with these regimens.
* Compare the overall survival of patients treated with these regimens.
* Characterize and contrast the adverse event and safety profile of these regimens in these patients.
* Compare the effects of these regimens on quality of life in these patients.

OUTLINE: This is a randomized, prospective, open-label, controlled, multicenter study. Patients are stratified according to study center, status of tumor (primary vs recurrent), carcinoma in situ (yes vs no), prior BCG therapy (yes vs no), and single dose of intravesical mitomycin C at the time of the most recent transurethral resection (yes vs no). Patients are randomized to 1 of 2 treatment arms.

* Arm I: Patients receive induction therapy comprising intravesical BCG once weekly for 6 weeks. Patients then receive maintenance therapy comprising intravesical BCG once weekly for 3 weeks.
* Arm II: Patients receive induction therapy comprising intravesical BCG once weekly for 6 weeks and oral gefitinib once daily for 12 weeks. Patients then receive maintenance therapy comprising intravesical BCG once weekly for 3 weeks and oral gefitinib once daily for 12 weeks.

In both arms, treatment with maintenance therapy repeats at 3, 6, 12, 18, 24, 30, and 36 months for a total of 7 courses in the absence of disease progression or unacceptable toxicity.

Quality of life is assessed at baseline, periodically during study therapy, and then at 3 and 6 months after completion of study therapy.

After study completion, patients are followed every 3 months for 2 years, every 6 months for 4 years, and then annually thereafter.

PROJECTED ACCRUAL: A total of 166 patients will be accrued for this study.

ELIGIBILITY:
DISEASE CHARACTERISTICS:

* Histologically confirmed transitional cell carcinoma (TCC) of the bladder meeting ≥ 1 of the following criteria:

  * Noninvasive papillary carcinoma (Ta) with ≥ 1 of the following characteristics:

    * Recurrence of bladder tumor(s) ≥ grade 2 within 6 months after transurethral resection (TUR)
    * Three or more bladder tumors ≥ grade 2 at the time of TUR
    * Bladder tumor(s) ≥ 5 cm in size and ≥ grade 2 at the time of TUR
    * Any grade 3 bladder tumor(s)
  * Carcinoma in situ (Tis)
  * At least grade 2 tumor that invades the subepithelial connective tissue (T1)
* Has undergone TUR of all visible bladder lesions within the past 21 to 60 days with biopsy of the underlying bladder wall for all tumors and cold-cup biopsy of all suspicious areas
* No metastatic disease as confirmed by negative radiology within the past 16 weeks, including the following:

  * Chest x-ray
  * Imaging of the upper urinary tract by 1 of the following methods:

    * CT scan, MRI, or ultrasound of the abdomen and pelvis
    * Intravenous pyelogram
    * Retrograde pyelogram
* No evidence of TCC of the upper urinary tract
* No mixed histology of bladder cancer (i.e., TCC and squamous cell carcinoma of the bladder or TCC and small cell carcinoma of the bladder) at the most recent TUR

PATIENT CHARACTERISTICS:

* ECOG performance status 0-2
* Life expectancy > 5 years
* Negative routine urine microscopy and negative urine culture within the past 14 days
* Willing to complete quality of life questionnaires in English or French

  * Inability to complete questionnaires due to illiteracy in English or French, loss of sight, or other reason allowed
* WBC ≥ 3,000/mm³
* Absolute neutrophil count ≥ 1,500/mm³
* Platelet count ≥ 100,000/mm³
* Bilirubin ≤ 1.5 times upper limit of normal (ULN)
* AST and ALT ≤ 1.5 times ULN
* Alkaline phosphatase ≤ 1.5 times ULN
* Creatinine ≤ 1.5 times ULN
* Not pregnant or nursing
* Negative pregnancy test
* Fertile patients must use effective contraception during and for 3 months after study completion
* No significant history of cardiac disease including, but not limited to, any of the following:

  * Uncontrolled high blood pressure
  * Unstable angina
  * Congestive heart failure
  * Myocardial infarction within the past year
  * Cardiac ventricular arrhythmias requiring medication
* No active urinary tract infection
* No active infection, including tuberculosis
* No serious underlying medical conditions that would impair the ability of the patient to receive protocol treatment
* No febrile illness or gross hematuria
* No impaired immune response from any cause (congenital, therapy, or disease)
* No clinically significant or untreated ophthalmologic condition (e.g., Sjögren's syndrome)
* No gastrointestinal conditions (e.g., Crohn's disease or ulcerative colitis)
* No history of psychiatric or neurological disorder that would limit study compliance
* No other malignancies except for adequately treated nonmelanoma skin cancer, curatively treated in situ cancer of the cervix, or other solid tumors curatively treated with no evidence of disease for ≥ 5 years
* No contraindications to spinal or general anesthesia as required for a TUR
* No known hypersensitivity to BCG or gefitinib
* No history of allergic reactions attributed to compounds of similar chemical or biologic composition to the study drugs

PRIOR CONCURRENT THERAPY:

* See Disease Characteristics
* More than 12 months since prior intravesical immunotherapy (including BCG +/- interferon)
* More than 6 months since prior intravesical chemotherapy (including mitomycin C, thiotepa, doxorubicin hydrochloride)

  * Single dose of intravesical mitomycin C at the time of the most recent TUR (within the past 21 to 60 days) allowed if considered standard care
* No other prior or concurrent immune modulator therapy
* No prior pelvic radiation
* No prior gefitinib
* No other concurrent experimental anticancer drugs
* No concurrent use of drugs that induce CYP3A4 enzymes that have been shown to significantly reduce plasma concentrations of gefitinib (including phenytoin, carbamazepine, barbiturates, rifampin, or Hypericum perforatum [St. John's wort])
* No concurrent grapefruit juice

Ages: 18 Years to 120 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 41 (Actual)
Dates: Start 2007-01-04 (Actual); Primary Completion 2012-01-06 (Actual); Study Completion 2012-01-06 (Actual)

PRIMARY OUTCOMES:
Time to treatment failure | 5 years

SECONDARY OUTCOMES:
Complete response rate in patients with carcinoma in situ | 5 years
Time to recurrence | 5 years
Time to progression | 5 years
Overall survival | 5 years
Adverse event and safety profile | 5 years
Quality of life | 5 years

CONTACTS AND LOCATIONS:
Overall Officials: Louis Lacombe, MD, Study Chair — Centre Hospitalier Universitaire de Quebec
Locations (6):
- Canada (6):
  - Clinical Research Unit at Vancouver Coastal, Vancouver, British Columbia
  - Hamilton and District Urology Association, Hamilton, Ontario
  - London Regional Cancer Program, London, Ontario
  - Univ. Health Network-Princess Margaret Hospital, Toronto, Ontario
  - CHUQ-Pavillon Hotel-Dieu de Quebec, Québec, Quebec
  - Centre hospitalier universitaire de Sherbrooke, Sherbrooke, Quebec

IPD SHARING:
Plan to Share IPD: No